CLINICAL TRIAL: NCT03241563
Title: A Randomized, Double-blind Comparison Trial of Subcutaneous Sodium Deoxycholate Injections With or Without Triamcinolone for Reduction of Submental Fat
Brief Title: Subcutaneous Sodium Deoxycholate Injections With or Without Triamcinolone for Reduction of Submental Fat
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATX-TRIAM-2016
Record Dates: First submitted 2017-03-02; First posted 2017-08-07 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Fat Reduction
MeSH Terms: interventions — Deoxycholic Acid; Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- without triamcinolone (Active Comparator): sodium Deoxycholate without triamcinolone
  Interventions: Drug: Sodium Deoxycholate
- with triamcinolone (Active Comparator): sodium Deoxycholate with triamcinolone
  Interventions: Drug: Sodium Deoxycholate; Drug: Triamcinolone

INTERVENTIONS:
Drug: Sodium Deoxycholate
  Other Names: Kybella
Drug: Triamcinolone — Triamcinolone 40mg/ml
  Arms: with triamcinolone

SUMMARY:
The subjects and evaluating investigator will be blinded to the treatment, thus maintaining double-blind status. By nature of the varying volumes of injection, the treating investigator will be unblinded to the treatment. A series of 3 injection sessions will be performed spaced 4 weeks apart.

Canfield Vectra 3D imaging will be performed at baseline and at each follow up visit. Follow up visits will be performed 3 and 5 days after each injection session to assess for side effect and tolerability profile. After the final injection session, additional follow up visits will be performed at days 90 and 180 to assess for efficacy. Subject weight will be recorded at baseline and at end of study.

DETAILED DESCRIPTION:
This is a Single-site randomized, double-blind comparison trial of Kybella injections with or without triamcinolone acetate for the reduction of submental fat. 20 subjects will be enrolled into the trial. Of these 20 subjects, 5 will be randomized to receive Kybella injections alone whereas 15 will receive Kybella plus triamcinolone acetate in the following way:

1. Kybella alone: 2 mg/cm2 of Kybella will be delivered in up to 50 injections spaced 1.0 cm apart at 0.2 mL/injection for a total dose of up to 100 mg of sodium deoxycholate.
2. Kybella plus triamcinolone: 0.2 mL of 2 mg/cm2 of Kybella will be mixed with 0.05 mL of 40 mg/mL of triamcinolone acetate and then delivered in up to 50 injections spaced 1.0 cm apart at 0.25 mL/injection for a total dose of up to 100 mg of sodium deoxycholate using a 30 gauge (or smaller) 0.5-inch needle.

The treatment area will be bounded superiorly by a line 1 cm inferior to the mandibular margin, laterally by the sternocleidomastoid muscles, and inferiorly by the hyoid bone. The subjects and evaluating investigator will be blinded to the treatment, thus maintaining double-blind status. By nature of the varying volumes of injection, the treating investigator will be unblinded to the treatment. A series of 3 injection sessions will be performed spaced 4 weeks apart.

Canfield Vectra 3D imaging will be performed at baseline and at each follow up visit. Follow up visits will be performed 3 and 5 days after each injection session to assess for side effect and tolerability profile. After the final injection session, additional follow up visits will be performed at days 90 and 180 to assess for efficacy. Subject weight will be recorded at baseline and at end of study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Females or Males in good general health age 18 - 65 years of age
* 2. Fitzpatrick skin types I-VI
* 3. Must be willing to give and sign a HIPPA form and informed consent form
* 4. Must be willing and able to comply with all study protocols and schedules
* 5. Must have submental fat graded by the investigator as 2 or 3 using the Clinician-Reported Submental Fat Rating Scale (PR-SMFRS)
* 6. Negative urine pregnancy test prior to each treatment (if applicable)
* 7. Female patients will be either of non-childbearing potential defined as: 7.1 Having no uterus 7.2 No menses for at least 12 months. Or; (WOCBP) women of childbearing potential must agree to use an effective method of birth control during the course of the study, such as: 7.3 Oral contraceptive pill, injection, implant, patch, vaginal ring, intrauterine device 7.4 Intrauterine coil 7.5 Bilateral tubal ligation 7.6 Barrier method used with an additional form of contraception (e.g., sponge, spermicide or condom) 7.7 Abstinence (If practicing abstinence must agree to use barrier method described above (7.6) if becomes sexually active) 7.8 Vasectomized partner (must agree to use barrier method described above (7.6) if becomes sexually active with unvasectomized partner)
* 8. Males must be willing to be clean shaven for all study visits
* 9. The patient must have had a stable weight (no fluctuation of >15 pounds in a year), diet, and physical activity for the previous 6 months

Exclusion Criteria:

* 1. Pregnancy, currently breast feeding or planning pregnancy for the duration of the trial
* 2. Any UNCONTROLLED systemic disease -a potential patient in whom therapy for a systemic disease is not yet stabilized will not be considered for entry into the study
* 3. Treatment with botulinum toxin injections in the neck or chin area within 6 months before randomization
* 4. Any Scars, unshaven hair, tattoos or jewelry on or near the proposed treatment area
* 5. Significant history or current evidence of a medical, psychological or other disorder that, in the investigator's opinion, would preclude enrollment into the study
* 6. An active dermatitis or open wound in the proposed treatment area
* 7. An active bacterial, fungal, or viral infection in the proposed treatment area
* 8. Pre-existing skin condition to the submental region that may confound evaluation or analysis, at investigator discretion
* 9. Previously treated with subcutaneous sodium deoxycholate to the submental region
* 10. Previously treated with focused ultrasound, radiofrequency, cryolipolysis or liposuction to the submental region within the previous 6 months
* 11. Any other laser, light energy device, or chemical peel treatment to the submental region within the previous 3 months
* 12. Pre-existing neurological or gastrointestinal condition leading to dysphagia, dysphonia or facial nerve palsy
* 13. Pre-existing medical condition other than increased submental fat that may result in increased submental fullness such as but not limited to thyroid enlargement, goiter, cervical lymphadenopathy etc., at investigator discretion
* 14. Must not have a planned fat reduction procedure of any variety to the submental region for the duration of the study
* 15. Must not have planned significant alterations in diet or physical activity that may result in significant fluctuations in weight
* 16. Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-04; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of Efficacy of Kybella with Triamcinolone in the Reduction of Submental Fat | 6 Months
  evaluate the efficacy associated with Kybella injections for the reduction of fat of the upper neck in the treatment of submental fat with and without added triamcinolone acetonide. An evaluator blinded to the study will grade the level of improvement of the submental fat using the Clinician Graded Submental Fat Rating Scale.

SECONDARY OUTCOMES:
Evaluation of Safety of Kybella with Triamcinolone for Reduction of Submental Fat | 6 months
  Differences in rates of edema, erythema, tenderness, and erosion/ulceration, based on blinded evaluator assessment, will be compared between subjects treated with Kybella with and without triamcinolone

CONTACTS AND LOCATIONS:
Overall Officials: Mitchel P Goldman, MD, Principal Investigator — DCLA
Locations (1):
- Dermatology Cosmetic Laser Medical Associates of La Jolla, Inc., San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No